CLINICAL TRIAL: NCT05301634
Title: Comparison Between Hemodynamic Effect of Bilateral Infraorbital Block Versus Intranasal Application of Bupivacaine in Patients Undergoing Transsphenoidal Pituitary Adenoma Resection.A Comparative Randomized Controlled Study
Brief Title: Comparison Between Bilateral Infraorbital Block Versus Intranasal Bupivacaine in Transsphenoidal Pituitary Adenoma Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdElKhalik Mahmoud Shaban, Lecturer of anaesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-532-2021
Record Dates: First submitted 2022-03-20; First posted 2022-03-31 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2022-05

CONDITIONS: Intraoperative Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): the patients will receive bilateral infraorbital block
  Interventions: Procedure: infraorbital block
- Group B (Active Comparator): the patients will receive topical intranasal application of bupivacaine
  Interventions: Procedure: topical intranasal bupivacaine

INTERVENTIONS:
Procedure: infraorbital block — the patients will receive bilateral infraorbital block
  Arms: Group A
Procedure: topical intranasal bupivacaine — the patients will receive topical intranasal application of bupivacaine
  Arms: Group B

SUMMARY:
The study will evaluate the efficacy of bilateral infraorbital nerve block versus preoperative nasal packing with long-acting local anesthetic bupivacaine in term of maintaining hemodynamics intraoperative within 20% below baseline to achieve adequate hypotensive anesthesia and longer duration of postoperative analgesia up to 24 hours in patients undergoing transsphenoidal pituitary adenoma resection.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II or III
* patients scheduled to undergo endoscopic transsphenoidal approach to remove tumor under general anesthesia

Exclusion Criteria:

* Patient's refusal
* Allergy to local anesthetics.
* Preoperative cerebrospinal fluid leak.
* Preoperative cardiac arrythmias.
* Seizure disorders.
* Patients with severe endocrinal disorders that affecting the craniofacial morphology as acromegaly and cushinoid features.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-02 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Mean arterial blood pressure | at the time of mucosal dissection

SECONDARY OUTCOMES:
Intraoperative need for magnesium sulphate | the entire duration of surgery
  Intraoperative need for iv magnesium sulphate up to 3 mg to maintain blood pressure 20% below baseline
Intraoperative need for fentanyl | the entire duration of surgery
  Intraoperative need for iv fentanyl blouses 0.5 μg/kg (maximum total dose 5 μg/kg for the entire procedure) if no response to magnesium sulphate
Intraoperative need for nitroglycerine | the entire duration of surgery
  Intraoperative need for iv nitroglycerine infusion (5 - 100 mic/min iv) if no response to magnesium sulphate and fentanyl
Postoperative need of pethidine | 24 hours postoprative
  Postoperative need of pethidine boluses 25 mg with max.100 mg
Postoperative pain assessed by Numeric pain score | 24 hours postoprative
  Pain score will be assessed postoperatively (using the verbal Numeric Rating Scale [NRS] 0-100; 0 = Non ,100 = Worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini hospital, Cairo, Egypt